CLINICAL TRIAL: NCT03123354
Title: Calibration and Validation of Masimo's O3 Regional Oximetry Device in Neonates, Infants and Children Undergoing Cardiac Catherization
Brief Title: Calibration and Validation of Masimo's O3 Regional Oximetry Device in Neonates, Infants and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RAMA0003
Record Dates: First submitted 2017-04-14; First posted 2017-04-21 (Actual); Results first posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test group (Experimental): All subjects are enrolled in the test group and receive an O3 regional oximeter sensor during their scheduled, general cardiac catheterization procedure.
  Interventions: Device: O3 regional oximeter sensor

INTERVENTIONS:
Device: O3 regional oximeter sensor — Noninvasive sensor that is placed on the forehead for measurement of oxygenation in the area under the sensor

SUMMARY:
The study will collect cerebral oximetry data from pediatric and neonatal subjects using the Masimo O3 regional oximetry device, for the purposes of device calibration and validation.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing cardiac catheterization procedure for treatment or diagnosis of cardiovascular disease
* 1 day to less than 18 years of age
* Weight between 3.5 and 40 kg
* Parental or legal guardian consent and subject assent

Exclusion Criteria:

* Failure to obtain written consent
* Equal or more than 18 years in age
* Weight more than 40kg or less than 3.5kg
* Jaundice with bilirubin levels higher than the reference range
* Subject has skin abnormalities affecting the digits such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown, nail polish or acrylic nails that would prevent motioning of SpO2 levels during the study or placement of cerebral oximeter

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- O3 Regional Oximeter Sensors: All subjects are enrolled in the test group and receive O3 regional oximeter sensors during their scheduled, general cardiac catheterization procedure.
  O3 regional oximeter sensors: Noninvasive sensors are placed on the forehead for measurement of oxygenation in the area under the sensor
Period: Overall Study
Arm/Group | O3 Regional Oximeter Sensors
Started | 44
Completed | 38
Not Completed | 6
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Population: The subjects included for the analysis are within the desired calibration range, with no sensor placement issues in the data collection time period.
Groups:
- O3 Regional Oximeter Sensors: All subjects are enrolled in the test group and receive the O3 regional oximeter sensor during their scheduled, general cardiac catheterization procedure.
  O3 regional oximeter sensor: Noninvasive sensors are placed on the forehead for measurement of oxygenation in the area under the sensor.
Arm/Group | O3 Regional Oximeter Sensors
Number analyzed (Participants) | 33
Age, Customized [Count of Participants; unit: Participants]
  0-23 months | 14
  2-12 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 16
  Ethnicity: Hispanic/Latino | 11
  Ethnicity: Asian | 4
  Ethnicity: Not Hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor by Arms Calculation of Percent rSO2
Description: The continuous measurements of regional oxygen saturation (rSO2) was compared against its reference cerebral oxygen saturation which is measured by a combination of arterial and jugular venous blood oxygen saturation. Absolute accuracy was determined by the root-mean-squared error (Arms). The Arms error value is calculated as the square root of the sum of the squares of mean bias and estimated standard deviation of bias. The bias is defined as the difference of the rSO2 and its blood reference.
Time Frame: One visit; up to 4 hours
Measure: Number; unit: %rSO2
Groups:
- O3 Regional Oximeter Sensors (Test Group): All pediatric subjects are enrolled in the test group and receive an O3 regional oximeter sensor during their scheduled, general cardiac catheterization procedure.
  O3 regional oximeter sensor: Noninvasive sensor that is placed on the forehead for measurement of oxygenation in the area under the sensor
Arm/Group | O3 Regional Oximeter Sensors (Test Group)
Number analyzed (Participants) | 33
%rSO2 | 5.0

ADVERSE EVENTS:
Time Frame: For each subject, adverse event data were collected up to 2 days after subject's single visit participation in the study.
Description: Subjects were observed during the procedure, as well as contacted via phone call up to 2 days after the procedure to gather adverse event information.
Groups:
- O3 Regional Oximeter Sensors: All subjects are enrolled in the test group and receive an O3 regional oximeter sensor during their scheduled, general cardiac catheterization procedure.
  O3 regional oximeter sensor: Noninvasive sensor that is placed on the forehead for measurement of oxygenation in the area under the sensor
Arm/Group | O3 Regional Oximeter Sensors
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 2/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | O3 Regional Oximeter Sensors (N=44)
Mild rash, localized to sensor location (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2014-12-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT03123354/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT03123354/SAP_001.pdf